CLINICAL TRIAL: NCT04522960
Title: Melatonin in Alzheimer's Disease: Effect on Disease Progression and Epileptiform Activity.
Acronym: MADE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UZB-NEU-002
Record Dates: First submitted 2020-08-13; First posted 2020-08-21 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Spinal Puncture; Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with dementia or mild cognitive impairment due to AD (Experimental): Dementia or MCI due to AD according to NIA-AA research criteria.
  Interventions: Diagnostic Test: MEG+hdEEG+MRI
- Healthy volunteers (Active Comparator): Age-and-gender matched healthy controls.
  Interventions: Diagnostic Test: MEG+hdEEG+MRI

INTERVENTIONS:
Diagnostic Test: MEG+hdEEG+MRI — We will perform several tests:
  * Neuropsychological testing to evaluate evolution of cognition during our study.
  * Lumbar puncture, blood sampling, saliva and urine collection to assess melatonin levels at several timepoints within these biological fluids.
  * MEG+hdEEG and MRI (to project MEG information) ; LTM-EEG to detect epileptiform activity in patients and healthy controls
  Other Names: Lumbar puncture; Long-term EEG monitoring; Blood sampling; Saliva collection; Urine collection; Neuropsychological examination

SUMMARY:
This is a long-term, prospective, observational study to investigate and compare the levels and rhythm of melatonin in patients with AD dementia, mild cognitive impairment due to AD and healthy volunteers. The investigators would like to validate the use of salivary and urine melatonin measurements as an alternative for blood/CSF melatonin. Furthermore, the investigators would like to assess the effects of melatonin levels on cognition by correlating the levels and changes on cognitive tasks over a two year time frame. The investigators will also investigate whether these effects could be due to its anticonvulsive properties.

DETAILED DESCRIPTION:
Melatonin production gets disrupted in AD, as shown in post-mortem pineal glands and CSF of AD patients. CSF melatonin levels are known to significantly drop in patients with Alzheimer's dementia. It is known that CSF melatonin levels are much higher than blood melatonin levels, due to melatonin secretion from the pineal recess directly into the third ventricle. It has never been investigated whether blood melatonin accurately correlates with CSF melatonin in AD, nor whether saliva or urine melatonin levels accurately reflect blood/CSF melatonin in the AD continuum. The investigators want to validate the use of blood, saliva and urine melatonin levels as alternative for CSF melatonin in the AD continuum to pave the way for further use of less invasive collection techniques (blood, saliva, urine instead of CSF) and to possibly study circadian rhythm in a less disrupting, in home environment (saliva, urine).

Furhtermore, melatonin exerts several potential anti-AD properties, including anti-inflammatory, anti-oxidant, tilting APP processing towards the non-amyloidogenic pathway, exerting positive effects on sleep and so on. In vivo studies furthermore point to anticonvulsive and antiepileptic effects of melatonin in a whole range of rodent models. Some evidence exists for a role of melatonin in prevention of epileptic seizures in humans.

The investigators want to investigate influence of melatonin on changes in cognition in a longitudinal way, and investigate influence on (sub)clinical epileptiform activity.

ELIGIBILITY:
Inclusion Criteria:

1. Dementia due to AD, according to National Institute on Aging-Alzheimer's Association (NIA-AA) criteria
2. MCI due to AD, according to NIA-AA criteria
3. Healthy controls: Age- and gender matched healthy controls

Exclusion Criteria:

Patients (AD dementia, MCI)

* Age < 18 years old
* Pregnancy
* Expected death due to illness within 2 years
* Pacemaker or other ferrromagnetic material that is not MRI compatible
* Other neurodegenerative or cerebrovascular disease
* Pattern compatible with NPH (clinically, imaging)
* Epilepsy
* Multiple sclerosis or other demyelinating disease
* Depression, psychosis or other mental disease
* Use of anti-epileptic drugs
* Alcohol or substance abuse
* Korsakoff syndrome
* Symptomatic liver disease
* Uncontrolled thyroid disorders
* Untreated HIV or syphilis
* Clinically significant vitamin B12 deficiency
* Severe systemic medical illness (eg end-stage cardiac disease, …)
* Use of melatonin, agomelatine, or other sleep medications
* Night worker
* REM sleep behavior disorder, OSAS

Healthy controls

* Age < 18 years old
* Pregnancy
* Pacemaker or other ferromagnetic material that is not MRI compatible
* Mild cognitive impairment or dementia of any cause
* Epilepsy
* Multiple sclerosis or other demyelinating disease
* Depression, psychosis or other mental disease
* Use of anti-epileptic drugs
* Alcohol or substance abuse
* Symptomatic liver disease
* Uncontrolled thyroid disorders
* Untreated HIV or syphilis
* Clinically significant vitamin B12 deficiency
* Severe systemic medical illness (eg end-stage cardiac disease, …)
* Use of melatonin, agomelatine, or other sleep medications
* Night worker
* REM sleep behavior disorder, OSAS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
CSF and blood melatonin levels in patients with AD dementia, MCI due to AD and healthy volunteers | 24 hours
  Comparison of CSF and blood melatonin levels between patients with MCI and dementia due to AD and healthy volunteers.
Blood, saliva and urine melatonin correlations | 24 hours
  Correlation between blood melatonin and urinary and salivary melatonin in the AD continuum
Melatonin influence on cognition | 2 years
  Correlations between melatonin levels and cognitive performance over a 2 year time frame. This will be assessed by use of neuropsychological testing including MMSE, MoCA, RBANS, VAT, ...
Melatonin influence on epileptiform activity | 8 weeks
  Correlations between melatonin levels and (subclinical) epileptiform activity. Over a time frame of 8 weeks patients will undergo neuropsychological testing (with MMSE, MoCA, RBANS, VAT...), LTM-EEG monitoring (during 24 hours), MEG + hdEEG.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No